CLINICAL TRIAL: NCT05837286
Title: Conservative Treatment of Trigger Finger: Outcomes of a Randomized Controlled Trial
Brief Title: Conservative Treatment of Trigger Finger
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Pamela Roberts, Executive Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00002410
Record Dates: First submitted 2023-04-05; First posted 2023-05-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Hand Injuries; Trigger Finger
MeSH Terms: conditions — Hand Injuries; Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: The primary objective of this study is to analyze the effectiveness of a nighttime PIP joint extension orthosis to improve pain and restore functional outcomes in TF and comparing two groups of participants with TF, one group receiving a cortisone injection only and the experimental group receiving the nighttime orthosis after cortisone injection using the QuickDASH.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group with Cortisone Injection of affected digit(s) and nighttime orthosis (Experimental): The experimental group will consist of receiving a PIP joint on the day they receive their cortisone injection. The Oval-8 ® will be issued to the subject by an Occupational Therapist to ensure correct fit and comfort as well as given written instructions for night use. The orthosis will be worn at night for 6-week duration. Participants will have 1 follow up phone call or email at the 6-week mark and then 1 follow up phone call or email at the 12 week mark by a member of the research team from the time they received their cortisone injection where the time for resolution of trigger finger symptoms, VAS (Visual Analogue Scale), subjective questionnaire and QuickDASH scores will all be recorded in their medical research file.
  Interventions: Device: Oval-8 ® Orthosis
- Control Group-No Orthosis (Active Comparator): The control group will be identical to the experimental group except without the use of a nighttime orthosis. Participants will have 1 follow up phone call or email at the 6-week mark and then 1 follow up phone call or email at the 12 week mark by a member of the research team from the time they received their cortisone injection where the time for resolution of trigger finger symptoms, VAS (Visual Analogue Scale), subjective questionnaire and QuickDASH scores will all be recorded in their medical research file.
  Interventions: Other: Cortisone injection only

INTERVENTIONS:
Device: Oval-8 ® Orthosis — The experimental group will consist of receiving a PIP joint on the day they receive their cortisone injection. The Oval-8 ® will be issued to the subject by an Occupational Therapist to ensure correct fit and comfort as well as given written instructions for night use. The orthosis will be worn at night for 6-week duration. Participants will have 1 follow up phone call or email at the 6-week mark and then 1 follow up phone call or email at the 12 week mark by a member of the research team from the time they received their cortisone injection where the time for resolution of trigger finger symptoms, VAS (Visual Analogue Scale), subjective questionnaire and QuickDASH scores will all be recorded in their medical research file.
  Other Names: Cortisone Injection
  Arms: Experimental Group with Cortisone Injection of affected digit(s) and nighttime orthosis
Other: Cortisone injection only — The control group will receive a cortisone injection and be instructed to move their fingers normally
  Arms: Control Group-No Orthosis

SUMMARY:
This study is to analyze the effectiveness of a nighttime extension orthosis after receiving a cortisone injection for the treatment of trigger finger to improve pain and restore functional outcomes. The investigators hypothesize that the extension orthosis will improve pain and functional outcomes compared to those without a digital night extension orthosis in those with trigger finger at 12 weeks from the injection.

DETAILED DESCRIPTION:
The purpose of the research is to analyze the effectiveness of a proximal interphalangeal joint (PIPJ) extension night orthosis status-post cortisone injection of the first annular pulley for the treatment of trigger finger to improve pain and restore functional outcomes. The investigators hypothesize that the extension orthosis will improve pain and functional outcomes (Quick Dash score) compared to those without a digital night extension orthosis in those with trigger finger at 12 weeks from the injection.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included
* Patients with trigger finger, aka stenosing flexor tenosynovitis
* Status post receiving cortisone injection of the affected digit(s)

Exclusion Criteria:

* Any records flagged with break the glass or research opt out
* Patients with rheumatoid arthritis
* Patients with a history of traumatic injury to the hand
* Cognitive or behavioral problems which would preclude informed consent
* Unable to speak and understand English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of Trigger Finger Symptoms | 6 Weeks
  Questionnaire used to determine resolution of Trigger Finger Symptoms
Resolution of Trigger Finger Symptoms | 12 Weeks
  Questionnaire used to determine resolution of Trigger Finger Symptoms

SECONDARY OUTCOMES:
Change in Pain | 6 weeks
  Visual Analogue Scale for Pain (0 pain free to 10 severe pain)
Change in Pain | 12 weeks
  Visual Analogue Scale for Pain (0 pain free to 10 severe pain)
Change in Perception of Function | 12 weeks
  QuickDash scores (0% no functional limitations to 100% disabled)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center Outpatient Rehabilitation Hand Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available for sharing.